CLINICAL TRIAL: NCT01829373
Title: Lung Cancer Immunotherapy With Vaccine 1650-G and Yeast Derived β-Glucan
Brief Title: Lung Cancer Vaccine Plus Oral Dietary Supplement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edward Hirschowitz (Other)
Collaborators: University of Louisville (Other)
Responsible Party: Sponsor-Investigator, Edward Hirschowitz, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG1006
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Vaccines; beta-Glucans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine plus oral beta glucan (Experimental): Vaccine plus oral beta glucan
  Interventions: Biological: vaccine 1650-G

INTERVENTIONS:
Biological: vaccine 1650-G
  Other Names: Beta Glucan capsule

SUMMARY:
This study tests the ability of the allogeneic cellular vaccine 1650-G vaccine to enhance immune recognition of tumor cells in patients with lung cancer. The vaccine is combined with an oral medication called beta glucan, an over the counter oral dietary supplement that may also stimulate the immune system in ways that helps the body eradicate cancer cells and reduce risk of recurrent cancer. The primary purpose of this study is to measure the changes in the number of immune cells that might help lower risk of cancer recurrence. The investigators do not yet know if the vaccine is effective in fighting cancer and will not know at the end of this study whether this has been of benefit.

DETAILED DESCRIPTION:
Open-label pilot (Phase II) study to assess the immunologic activity of a cellular vaccine composed of killed allogeneic tumor cells (1650-G) and GM-CSF in patients with stage I-IIIA NSCLC after definitive therapy. (Surgery, Surgery plus Radiation Therapy, or Surgery, Radiation Therapy plus Adjuvant Chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, surgically resected stage I-IIIA NSCLC (Bronchoalveolar carcinomas are eligible).
* Must have read, voiced understanding of and signed an informed consent document.
* At least 21 years old
* At least 4 weeks but no more than 12 months post surgical resection.
* At least 4 weeks since completion of chemotherapy or radiation therapy (adjuvant)
* No evidence of disease following definitive initial therapy evidenced by a CXR, CT or PET scan within 6 weeks of accrual.
* ECOG performance status of 0 to 2 (Section 19.1)
* Adequate organ and marrow function defined as follows:
* Hemoglobin ≥9.0 gm/dL
* Absolute neutrophil count (ANC) ≥1,500/mcl
* Platelet count ≥ 75,000/mcl
* AST <2.5 x upper limit of normal
* ALT <2.5 x upper limit of normal
* Creatinine Clearance (CCr) >50 ml/min
* Female patients must not be pregnant or breastfeeding. Women of childbearing potential must have a negative pregnancy test and agree to use acceptable birth control until the "analysis for immunologic response" 16 weeks after the second vaccination. Study doctor will discuss acceptable methods of contraception with patients.

Exclusion Criteria:

* Patients must not have not have no active residual or progressive lung cancer (Stable Disease)
* History of other malignancies unless they have had curative treatment completed greater than (≥) five years prior to enrollment or one of the following; appropriately managed Carcinoma in situ, basal cell carcinoma of the skin or non-metastatic squamous cell carcinoma of the skin.
* Patients must not be chronically immunosuppressed.
* Patients with HIV and other immunosuppressive disorders and patient who chronically use immunosuppressive medications are excluded. Patients should not be taking immuno-suppressive steroids for at least 4 weeks prior to enrollment
* Individuals with conditions that might require shorter courses of immunosuppressive oral medications (e.g. steroids) during the initial 16 weeks following immunization are excluded.
* Patients should not have taken or plan to take other immunologically active agents (eg flu vaccines) for a twelve week period, beginning 2 weeks prior to first dose of beta-glucan and two weeks following last dose of beta glucan.
* Patients must not have a known history of infectious hepatitis.
* Because of the unknown effects of this treatment on the fetus pregnant females, and childbearing females and males not willing to use contraception are not eligible.
* Patients must not have cardiovascular disease defined as:
* New York Heart Association Class III or IV congestive heart failure
* hemodynamically significant valvular heart disease
* myocardial infarction within the last six months
* active angina pectoris
* uncontrolled ventricular arrhythmias
* stroke within one year
* known cerebrovascular disease
* Patients may not have received any other investigational agents or participated in any investigational drug study within 4 weeks preceding initiation of study treatment.
* No known allergies or history of allergic reactions to any colony stimulating factor (GCSF, GMCSF)
* No known intolerance to yeast derive β-glucan

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Immunologic response to vaccine | 12 months
  Increase in number of peripheral blood T cells recognizing cancer antigens

CONTACTS AND LOCATIONS:
Overall Officials: Edward Hirschowitz, MD, Principal Investigator — University of Kentucky; John Yannelli, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Background] Hirschowitz EA, Mullins A, Prajapati D, Baeker T, Kloecker G, Foody T, Damron K, Love C, Yannelli JR. Pilot study of 1650-G: a simplified cellular vaccine for lung cancer. J Thorac Oncol. 2011 Jan;6(1):169-73. doi: 10.1097/JTO.0b013e3181fb5c22. PMID 21150468
- [Background] Hirschowitz EA, Foody T, Hidalgo GE, Yannelli JR. Immunization of NSCLC patients with antigen-pulsed immature autologous dendritic cells. Lung Cancer. 2007 Sep;57(3):365-72. doi: 10.1016/j.lungcan.2007.04.002. Epub 2007 May 16. PMID 17509725
- [Background] Hirschowitz EA, Foody T, Kryscio R, Dickson L, Sturgill J, Yannelli J. Autologous dendritic cell vaccines for non-small-cell lung cancer. J Clin Oncol. 2004 Jul 15;22(14):2808-15. doi: 10.1200/JCO.2004.01.074. PMID 15254048